CLINICAL TRIAL: NCT01429350
Title: The THERAPY Trial: The Randomized, Concurrent Controlled Trial to Assess the Penumbra System's Safety and Effectiveness in the Treatment of Acute Stroke
Brief Title: Assess the Penumbra System in the Treatment of Acute Stroke
Acronym: THERAPY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP 4338
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; acute intervention; thrombolysis; rtPA; internal carotid artery; middle cerebral artery; mechanical thrombectomy; Penumbra System; clot length; mRS; NIHSS
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV rtPA (Active Comparator): IV infusion of rtPA at 0.9mg/kg to a maximum of 90mg
  Interventions: Drug: intravenous (IV) recombinant human tissue plasminogen activator (rtPA)
- IV rtPA and IA Penumbra System (Experimental): Dual IV rtPA therapy (0.9mg/kg to a maximum of 90mg) and IA adjunctive treatment with the Penumbra System
  Interventions: Device: Penumbra System

INTERVENTIONS:
Drug: intravenous (IV) recombinant human tissue plasminogen activator (rtPA) — 0.9mg/kg to a maximum of 90mg
  Other Names: recombinant tissue plasminogen activator, Alteplase
  Arms: IV rtPA
Device: Penumbra System — The Penumbra System is an aspiration based mechanical thrombectomy device
  Arms: IV rtPA and IA Penumbra System

SUMMARY:
The purpose of this trial is to assess the safety and effectiveness of the Penumbra System as an adjunctive treatment to intravenous (IV) recombinant human tissue plasminogen activator (rtPA)in patients with acute ischemic stroke from large vessel occlusion in the brain. IV rtPA is the only drug approved for the treatment of acute ischemic stroke but it does not work very well in cases where the stroke is caused by a large vessel occlusion. The hypothesis being tested is to determine if the addition of a treatment by a mechanical thrombectomy device like the Penumbra System can improve the clinical outcome of the patient over just using IV rtPA alone.

DETAILED DESCRIPTION:
Current therapies for acute stroke are limited to the intravenous administration of a intravenous (IV) recombinant human tissue plasminogen activator (rtPA) for thrombolysis of the affected cerebral arteries within 3-4.5 hours from symptom onset, and the use of intra-arterial (IA) endovascular mechanical clot retrieval devices within 8 hours from ictus, all of which have limitations as mono therapies. For example, IV rtPA may not be very efficacious in large vessel occlusion and the long term effects of mechanical thrombectomy devices on patient functional outcome is unknown. This is a randomized, concurrent controlled study to assess the safety and effectiveness of the Penumbra System as adjunctive therapy to IV rtPA in the acute intervention of acute ischemic stroke. Patients presenting with symptoms of acute ischemic stroke who have evidence of a large clot burden (clot length > 8mm) in the anterior circulation will be assigned to either IV rtPA therapy alone (0.9mg/kg to a maximum of 90mg) or a combined IV rtPA therapy (0.9mg/kg to a maximum of 90mg) and intra-arterial (IA) adjunctive treatment with the Penumbra System. Each treated patient will be followed and assessed for 3 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. From 18 to 85 years of age
2. Present with symptoms consistent with an acute ischemic stroke and eligible for IV rtPA therapy (patients presenting 3-4.5 hrs from symptom onset are not eligible if they are >80 yrs of age, have a history of stroke and diabetes, anticoagulant use (even if INR is <1.7) and have a NIHSS score >25
3. Evidence of a large vessel occlusion in the anterior circulation with a clot length of 8mm or longer
4. NIH Stroke Scale (NIHSS) score 8 or greater or aphasic at presentation
5. Signed informed consent

Exclusion Criteria:

1. History of stroke in the past 3 months.
2. Females who are pregnant
3. Pre-existing neurological or psychiatric disease that could confound the study results such as a pre-stroke mRS score 1 or greater
4. Known severe allergy to contrast media
5. Uncontrolled hypertension (defined as systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg)
6. CT evidence of the following conditions at randomization:

   * Significant mass effect with midline shift
   * Any acute ischemic changes in >1/3 of the affected middle cerebral artery territory
   * Evidence of intracranial hemorrhage
7. Angiographic evidence of tantem extracranial occlusion or an arterial stenosis proximal to the occlusion that requires treatment prior to thrombus removal. Moderate stenosis not requiring treatment is not an exclusion
8. Angiographic evidence of preexisting arterial injury
9. Rapidly improving neurological status prior to randomization
10. Bilateral stroke
11. Intracranial tumors
12. Known history of cerebral aneurysm or arteriovenous malfunction
13. Known hemorrhagic diathesis, coagulation deficiency, or on anticoagulant therapy with an International Normalized Ratio (INR) of >1.7
14. Baseline platelets <50,000
15. Use of IV heparin in the past 48 hours with PPT >1.5 times the normalized ratio
16. Pre-treatment glucose <50mg/dL or >300mg/dL
17. Life expectancy less than 90 days prior to stroke onset
18. Participation in another clinical investigation that could confound the evaluation of the study device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, MS, Principal Investigator — Vanderbilt University Medical Center; Pooja Khatri, MD, Principal Investigator — Department of Neurology, University of Cincinnati; Osama Zaidat, MD, MSc, Principal Investigator — Neurointerventional Program, Medical College of Wisconsin
Locations (4):
- United States (4):
  - Endovascular Surgical Neuroradiology, Swedish Medical Center, Denver, Colorado
  - Department of Neurological Surgery, Gainesville, Florida
  - Neurosurgery, Rush University Medical Center, Chicago, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Yoo AJ, Khatri P, Mocco J, Zaidat OO, Gupta R, Frei D, Lopes D, Shownkeen H, Berkhemer OA, Meyer D, Hak SS, Kuo SS, Buell H, Bose A, Sit SP, von Kummer R; THERAPY Trial Investigators. Impact of Thrombus Length on Outcomes After Intra-Arterial Aspiration Thrombectomy in the THERAPY Trial. Stroke. 2017 Jul;48(7):1895-1900. doi: 10.1161/STROKEAHA.116.016253. Epub 2017 Jun 8. PMID 28596447

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System
Started | 53 | 55
As-Treated | 62 | 43
Per Protocol | 41 | 37
90 Day | 46 | 50
Completed | 46 | 50
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10) | 67 (11) | 68.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 51
  Male | 23 | 34 | 57

OUTCOME MEASURES:

1. Primary Outcome: Good Functional Outcome as Defined by a Modified Rankin Score of 0-2
Description: The assessor is blinded to patient treatment assignment.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System
Number analyzed (Participants) | 46 | 50
Participants | 14 | 19

2. Primary Outcome: Incidence of All Serious Adverse Events
Description: A Serious Adverse Event is defined as an event that:
  1. Led to death
  2. Led to a serious deterioration in the health of the patient that:
     * Resulted in life-threatening illness or injury
     * Resulted in permanent impairment of a body structure or a body function
     * Required in-patient hospitalization or prolongation of existing hospitalization
     * Resulted in medical or surgical intervention to arrest permanent impairment to body structure or a body function
     * Led to fetal distress, fetal death or a congenital abnormality or birth defect
Time Frame: 90 days
Population: The number of participants here are taken from the as-treated population, where IV tPA alone is 62 which differs from the number of initial participants started based on participant flow. This is due to 9 subjects who were randomized to Penumbra System receiving IV tPA Alone and no Penumbra System was used.
Measure: Count of Participants; unit: Participants
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System
Number analyzed (Participants) | 62 | 43
Participants | 30 | 18

3. Secondary Outcome: Good Clinical Outcome
Description: Good clinical outcome at 30 days post-procedure as defined by a 10 points or more improvement in the NIH stroke scale score at Discharge, a NIH stroke scale score of 0-1 at Discharge; or a 30-day modified Rankin scale score of 0-2
Time Frame: 30 days
Population: 30 day good clinical outcome based on ITT (intent-to-treat) population.
Measure: Count of Participants; unit: Participants
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System
Number analyzed (Participants) | 53 | 53
Participants | 17 | 24

4. Secondary Outcome: Incidence of Symptomatic and Asymptomatic Intracranial Hemorrhage
Description: A symptomatic intracranial hemorrhage is defined as 24 hour CT evidence of an ECASS defined ICH and a 4-point or more worsening of the NIH Stroke Scale score
Time Frame: 90 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System
Number analyzed (Participants) | 62 | 43
Participants | 6 | 4

ADVERSE EVENTS:
Description: The number of participants are taken from the as-treated population.
  Serious Adverse Events: The number of participants are taken from the as-treated population, where IV tPA alone is 62 which differs from the number of initial participants. This is due to 9 subjects who were randomized to Penumbra System receiving IV tPA Alone and no Penumbra System was used.
Arm/Group | IV rtPA | IV rtPA and IA Penumbra System
Serious Adverse Events (participants affected / at risk) | 32/62 | 20/43
Other Adverse Events (participants affected / at risk) | 58/62 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV rtPA (N=62) | IV rtPA and IA Penumbra System (N=43)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Hematemesis (Gastrointestinal disorders) | 2 | 1
Chest pain (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 3 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 1
Haemorrhage intracranial (Nervous system disorders) | 3 | 2
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV rtPA (N=62) | IV rtPA and IA Penumbra System (N=43)
Anaemia (Blood and lymphatic system disorders) | 4 | 8
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 4 | 1
Aortic valve sclerosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 11 | 10
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 4 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 2
Extrasystoles (Cardiac disorders) | 1 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 1
Left valve incomptence (Cardiac disorders) | 0 | 1
Left atrial dilatation (Cardiac disorders) | 0 | 1
Mitral valve calcification (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 3
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dry Eye (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 9 | 5
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Hematesis (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 1
Peptic ulcer (General disorders) | 1 | 0
Vomiting (General disorders) | 3 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 4 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 7 | 5
Thrombosis in device (General disorders) | 0 | 1
Unevaluable event (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 1
Vessel puncture site haemorrhage (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridal infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Eosophageal candiasis (Infections and infestations) | 0 | 1
Oral candiasis (Infections and infestations) | 3 | 1
Oral infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 16 | 12
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 3
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Antithrombin III decreased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 1
Troponin increased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hypovolaemia (General disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 5
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Aphasia (Nervous system disorders) | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 9 | 5
Carotid artery dissection (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Cerebral artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 7 | 1
Cerebrovascular spasm (Nervous system disorders) | 0 | 4
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 19 | 14
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 8 | 6
Hydrocephalus (Nervous system disorders) | 8 | 6
Hypertonia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 1
Intracranial pressure increased (Nervous system disorders) | 2 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 1
Stroke in evolution (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 3
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 7 | 5
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 0
Mental status changes (Psychiatric disorders) | 2 | 3
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Calculus urinary (Psychiatric disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3
Incontinence (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Reproductive system and breast disorders) | 0 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Accelerated hypertension (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 6
Hypotension (Vascular disorders) | 5 | 9
Orthostatic hypotension (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Vascular calcification (Vascular disorders) | 0 | 1
Vasospasm (Vascular disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days